CLINICAL TRIAL: NCT01523444
Title: Advancing Adolescent Screening and Brief Intervention Protocols in Primary Care Settings
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study not funded.
Sponsor: Treatment Research Institute (Other)
Responsible Party: Sponsor
Organization: Public Health Management Corporation (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASBIRT-PA-11-311
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Substance Abuse
Keywords: Adolescents; Screening; Advice; Referral
MeSH Terms: conditions — Substance-Related Disorders | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment as Usual (No Intervention)
- computer Screening & Brief Advice (Active Comparator): All participants receiving care at the site assigned to the computer-facilitated screening and brief advice (cSBA) condition will receive the cSBA intervention as part of their care at that clinic.
  Interventions: Behavioral: computer-assisted Screening & Brief Advice
- computer Screening & Brief Advice Plus (Experimental): All participants receiving care at the site assigned to the cSBA+ condition will receive the cSBA intervention elements plus the delivery of a brief, two-session motivational enhancement therapy (MET) intervention to be delivered a Behavioral Health Counselor (BHC) at the clinic immediately after meeting with the primary care provider as part of care at that clinic.
  Interventions: Behavioral: computer-assisted Screening & Brief Advice Plus

INTERVENTIONS:
Behavioral: computer-assisted Screening & Brief Advice — The computer-facilitated screening and brief advice (cSBA) intervention is a self-administered, computer-facilitated screening that asks about lifetime and past-12-month use of substances followed by scientific information about how substance use affects health and true-life stories illustrating the health risks of substance use. The cSBA program prints out a Report Form with the screening results, risk level, and "talking points" designed to prompt a 2 to 3-minute provider/teen conversation about the health effects of substance use, which recommends abstinence.
  Arms: computer Screening & Brief Advice
Behavioral: computer-assisted Screening & Brief Advice Plus — The cSBA+ intervention contains cSBA intervention elements plus the delivery of a brief, two-session motivational enhancement therapy (MET) intervention to be delivered a Behavioral Health Counselor (BHC) at the clinic immediately after meeting with the primary care provider. In the first session of this intervention, youth should be encouraged to think about: (1) The role alcohol and drugs play in his/her life; (2) His/her personal goals for changing alcohol and drug use; (3) Strategies for reaching and maintaining goals. The goal at the end of the session is positive movement in the direction of abstinence or change. The aim of the second session is reinforcement of goals set forth in the prior meeting with the BHC.
  Arms: computer Screening & Brief Advice Plus

SUMMARY:
This proposed study tests the effectiveness and examines the implementation of screening and brief intervention techniques to delay initiation and reduce substance use among adolescents accessing medical care in Federally Qualified Health Care settings with a computer-facilitated intervention. The primary hypothesis is that participants in the intervention groups will be more likely to cease or reduce substance use at follow-up compared to clients in the treatment as usual condition.

DETAILED DESCRIPTION:
The aims of the proposed 5-year study are threefold: (1) To examine the effectiveness of a computer-facilitated Screening and Brief Advice (cSBA) to reduce initiation and substance abuse among adolescents in a novel setting; (2) To examine the comparative effectiveness of adding a Brief Intervention and Referral to Treatment component to the cSBA intervention among adolescents in these centers; (3) To examine factors facilitating and inhibiting the implementation of SBIRT-type procedures with adolescents in FQHCs.

ELIGIBILITY:
Inclusion Criteria:

* 12-18 year old patients seeking care at the primary care participating sites

Exclusion Criteria:

* Unable to read and understand English
* Medically unstable
* Unavailable for follow-up

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2016-02 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Reduced substance use | 3 and 12 months

SECONDARY OUTCOMES:
Initiation of substance use | 3 and 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Amy Mericle, Ph.D., Principal Investigator — Treatment Research Institute
Locations (1):
- Treatment Research Institute, Philadelphia, Pennsylvania, United States